CLINICAL TRIAL: NCT04644432
Title: A Phase II Study of an Individualized Treatment Strategy for Patients With Metastatic Non-clear Cell Renal Cell Carcinoma
Brief Title: Individualized Treatment Strategy for Patients With Metastatic Non-clear Cell Renal Cell Carcinoma
Acronym: INDIGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Ida Rasmussen, Principal investigator, MD, Herlev and Gentofte Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UR1909; 2019-001316-38 (EudraCT Number); PACTIUS (Other: P-2019-232); GCP (Other: 2019-1153)
Record Dates: First submitted 2020-10-30; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Kidney Neoplasm; Urologic Neoplasms; Urogenital Neoplasms
Keywords: non-clear cell renal cell carcinoma; liquid biopsy; patient reported outcomes; gene expression
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A - for patients with a DNA mutation that match a targeted treatment (Experimental): Listed below are the possible study drugs and dosages:
  Erlotinib 150 mg once a day for 4 weeks.
  Osimertinib 80 mg once a day for 4 weeks.
  Alectinib 600 mg twice a day for 4 weeks
  Dabrafenib 150 mg twice a day combined with Trametinib 2 mg once a day for 4 weeks
  Trastuzumab-emtansin iv infusion 3.6 mg/kg every 3rd week
  Olaparib 400 mg twice a day for 4 weeks
  Pembrolizumab iv infusion 2 mg/kg every 3rd week
  Cabozantinib 60 mg once a day for 4 weeks
  Crizotinib 250 mg twice a day for 4 weeks
  Palbociclib 125 mg once a day in3 weeks, hereafter pause for one week
  Imatinib 400 mg once a day for 4 weeks
  If the patient can fit in several arms, arm A or the arm closest to arm A is chosen.
  Interventions: Drug: Medication (A specification is listed under each arm); Other: Patient reported outcomes measurement
- B - for patients with an angiogen profile (Experimental): Study drug: Sunitinib peroral tablet 50 mg once a day for 4 weeks, hereafter pause for 2 weeks (4/2 schedule or 2/1 schedule).
  If the patient can fit in several arms, arm A or the arm closest to arm A is chosen.
  Interventions: Drug: Medication (A specification is listed under each arm); Other: Patient reported outcomes measurement
- C - for patients with an immune profile (Experimental): Study drug: Nivolumab iv infusion 6 mg/kg (max 480 mg) every 4th week.
  If the patient can fit in several arms, arm A or the arm closest to arm A is chosen.
  Interventions: Drug: Medication (A specification is listed under each arm); Other: Patient reported outcomes measurement
- D - for patients that have neither mutations nor an immune- or angiogen profile (Experimental): Study drug: Nivolumab iv infusion 6 mg/kg (max 480 mg) every 4th week.
  If the patient can fit in several arms, arm A or the arm closest to arm A is chosen.
  Interventions: Drug: Medication (A specification is listed under each arm); Other: Patient reported outcomes measurement

INTERVENTIONS:
Drug: Medication (A specification is listed under each arm) — Study drugs and dosages are listed in the description of arms.
Other: Patient reported outcomes measurement — PRO questionnaires regarding symptoms and side effects with questions selected from the Nation Cancer Institute Patient Reported Outcomes-Common Terminology Criteria for Adverse Events.
  The patient receive individual advices according to the patient's answers to reduce the symptoms and side effects or is instructed to contact the hospital.
  For monitoring quality of life the EORTC QLQ-C30 is used. All questionnaires are in Danish.
  Other Names: PRO

SUMMARY:
The purpose of the open-label INDIGO-study is to examine whether a first line individualized treatment strategy based on DNA and RNA analyses from the patient's tumor is feasible. Moreover, to involve the patient further in their treatment via patient-reported outcomes (PRO) measurements in a value-based healthcare setup with simultaneous analyses of the financial costs of this strategy.

The patients are assigned into 4 treatment arms according to the results of their DNA and RNA analyses. All patients receive electronic questionnaires regarding symptoms and side effects weekly and questionnaires regarding quality of life monthly. Based on each patient's answers of the questionnaires the patient receives advices in the app to reduce the symptoms and side effects or the patient is instructed to contact the hospital.

The hypothesis: Basing the choice of first-line treatment for DNA mutations and RNA profiles in a heterogeneous patient population increases the overall response rate for the total population to 30% compared to 10% for historical cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained before any study-related procedures start.
2. The patient must be willing and able to follow the protocol.
3. Age ≥ 18 years
4. Histological biopsy-confirmed inoperable, locally advanced or metastatic non-cc RCC or 100% sarcomatoid tumour arising from the kidney found unsuited for surgery with a curative intent. Nephrectomy is not mandatory.

   1. If the primary disease was diagnosed more than 1 year ago, a fresh medium needle biopsy must be collected to confirm the diagnosis and tissue must be collected for DNA and RNA analyses.
   2. If a patient with inoperable relapse had a nephrectomy less than 1 year ago, and no tissue samples are stored in Dansk CancerBiobank, a fresh medium needle biopsy must be collected for DNA and RNA analyses.
   3. In cases where metastatic disease was confirmed by biopsy more than 1 year ago without initiated treatment, the patient is offered a fresh medium needle biopsy, but this is not mandatory for inclusion.
   4. If the patient had a nephrectomy using tissue from Dansk CancerBiobank and has been diagnosed with metastases within 1 year, the patient must be offered a fresh medium needle biopsy from a metastasis if the metastasis is easily accessible for biopsy, but a fresh biopsy is not mandatory for inclusion.
   5. A medium needle biopsy is mainly taken from a metastasis, but biopsy from a renal tumour is allowed.
   6. A biopsy may not be taken from bones as it cannot be used for molecular analysis.
   7. If the primary tumour is a proven clear cell RCC, but the biopsy from a metastasis shows non-cc RCC, the patient can be included in the study.
5. Sufficient tissue for DNA analyses, corresponding to 10 slides and RNA analyses corresponding to 1000 tumour cells.
6. Females with a negative pregnancy test or of non-childbearing potential (menopausal, hysterectomy or ovariectomy) and non-breastfeeding.
7. Females of childbearing potential (<2 years after last menstrual period) and males must use effective contraception (pills, intrauterine device, diaphragm or condom with spermicide or sterilisation).
8. Measurable disease (according to RECIST 1.1 criteria)
9. Karnofsky Performance status ≥ 70% / ECOG Performance status 0-2.
10. Life expectancy more than 3 months.
11. At baseline, the laboratory values must be: Haematology: Leukocytes ≥ 3.0 x 109/l, thrombocytes ≥ 100 x 109/l, haemoglobin ≥ 6.2 mmol/l.
12. Biochemistry: International Normalized Ratio (INR) ≤ 1.5, APTT ≤ 1.5 x upper limit of normal (ULN) Total bilirubin ≤ 1.5 x ULN, aspartate transaminase, alanine aminotransferase ≤ 2.5 x ULN for patients without liver metastases, ≤ 5 x ULN for patients with liver metastases. Estimated glomerular filtration rate (eGFR) > 30.

Exclusion Criteria:

1. Previous systemic treatment for metastatic RCC (including neoadjuvant treatment).
2. Former adjuvant treatment with immune checkpoint inhibitors.
3. Major surgical procedure, open surgical biopsy or significant trauma within 28 days prior to initiation.
4. Serious non-healing wound, ulcer or bone fracture.
5. Auto-immune disease or other condition requiring systemic treatment with either corticosteroids (prednisolone > 10 mg/day or similar) or other immunosuppressive drugs
6. Metastases in the central nervous system (CNS). The patient must have an MRI scan (preferred) or CT scan of the brain (using contrast agent if possible) within 28 prior to initiation.
7. Seizures which cannot be managed with standard medical treatment.
8. If urine dipstick with protein ≥ 3+, urine must be collected over a period of 24 hours which must be < 3.5 grams/day. If degree 2 proteinuria, urine must be collected over a period of 24 hours prior to each prescription.
9. Other malignancy within 5 years (except for curatively treated basal cell carcinoma of the skin and/or cervix carcinoma in situ).
10. Uncontrolled hypertension (≥ 150 mm Hg systolic and/or ≥ 100 mm Hg diastolic) despite maximum antihypertensive medical treatment.
11. Clinically significant (i.e. active) cardiovascular disease, such as cerebrovascular conditions (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) congestive heart failure ≥ degree III or serious cardiac arrhythmia requiring medical treatment. Patients with well-managed Atrial fibrillation/ atrial flutter may be included.
12. Treatment using other investigational drugs or participation in other studies.
13. Previous or current other diseases, metabolic dysfunction, clinical findings on physical examination or clinical laboratory findings that give suspicion of a disease or condition that would contraindicate the use of an investigational drug or a patient with a high risk of treatment complications.
14. Patients where the investigator finds that patient compliance prevents safe completion of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-09-06 (Estimated); Study Completion 2022-09-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 30 months
  The total share of patients who have received treatment with complete and partial response assessed radiologically based on RECIST v.1.1.
Time to treatment failure (TTF) | 30 months
  The time from start up day 1 until discontinuation of treatment, regardless of the reason.

SECONDARY OUTCOMES:
Overall Survival (OS) | 30 months
  Overall survival for the total population
Progression-Free Survival (PFS) | 30 months
  Progression-free survival for the total population
Disease Control Rate (DCR) | 30 months
  Disease control rate (complete response + partial response + stabile disease) for the total population based on RECIST v1.1 criteria
Response duration | 30 months
  Response duration for the total population.
Use of PRO tools | 30 months
  The patients' use of PRO tools during treatment assessed with the validated Patient Feedback Form
PRO and PRO-CTCAE | 30 months
  Number of and changes in Patient-reported outcomes according to PRO-CTCAE from baseline.
NCI-CTCAE | 30 months
  Number of and types of adverse events according to NCI-CTCAE
Hospital admissions | 30 months
  Number of hospital admissions

OTHER OUTCOMES:
Quality of life questionnaires EORTC QLQ-C30 (general quality of life questionnaire) | 36 months
  Changes in quality of life measured with EORTC-C30 every 4th week during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ida Marie L Rasmussen, MD, Principal Investigator — Department of Oncology, Herlev and Gentofte Hospital
Locations (1):
- Department of Oncology, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen IML, Soerensen AV, Moller AK, Persson GF, Palshof JA, Taarnhoj GA, Pappot H. Individualizing the Oncological Treatment of Patients With Metastatic Non-Clear Cell Renal Cell Carcinoma by Using Gene Sequencing and Patient-Reported Outcomes: Protocol for the INDIGO Study. JMIR Res Protoc. 2022 Sep 15;11(9):e36632. doi: 10.2196/36632. PMID 36107483